CLINICAL TRIAL: NCT06258720
Title: Interventional, Randomized, Open-label, Parallel-group, Single-dose Trial Investigating the Safety, Immunogenicity, Tolerability, and Pharmacokinetic Properties of Lu AF82422 in Healthy Chinese and Caucasian Participants
Brief Title: A Trial Investigating Lu AF82422 in Healthy Chinese and Caucasian Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19728A
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Healthy Participants
Keywords: Safety; Immunogenicity; Tolerability; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lu AF82422 Dose Level 1 (Experimental): Participants will receive a single intravenous (IV) infusion of Lu AF82422
  Interventions: Drug: Lu AF82422
- Lu AF82422 Dose Level 2 (Experimental): Participants will receive a single IV infusion of Lu AF82422
  Interventions: Drug: Lu AF82422

INTERVENTIONS:
Drug: Lu AF82422 — Lu AF82422 solution for intravenous infusion

SUMMARY:
The main goals of this trial are to learn more about a) the safety and tolerability of Lu AF82422 (any new or worsening medical issues the participants have with treatment), b) the immunogenicity of Lu AF82422 (the potential for the drug to trigger an unwanted immune response), and c) the pharmacokinetic parameters of Lu AF82422 (how the drug is absorbed, distributed, and processed by the body). During the trial, healthy adult Chinese and Caucasian participants will receive a single dose of Lu AF82422, which will be given as an intravenous infusion.

ELIGIBILITY:
Inclusion Criteria:

* For Chinese participants only: The participant is Chinese, defined as having four Chinese grandparents.
* For Caucasian participants only: The participant is Caucasian, defined as having four Caucasian grandparents.
* The participant has a Body Mass Index (BMI) ≥19 and ≤26 kilograms per square meter (kg/m2) at the Screening Visit and at the Baseline Visit.
* The participant is, in the opinion of the investigator, generally healthy based on medical history, a physical examination, a neurological examination, vital signs, an electrocardiogram (ECG), and the results of the clinical chemistry, haematology, urinalysis, serology, and other laboratory tests.

Exclusion Criteria:

* The participant has previously been enrolled in this trial.
* The participant has previously been dosed with Lu AF82422.
* The participant has participated in a clinical trial <30 days prior to the Screening Visit.
* The participant has taken any investigational medicinal product <3 months or <5 half-lives of that product, whichever is longer, prior to administration of the IMP.
* The participant is pregnant, breastfeeding, intends to become pregnant, or is of childbearing potential and not willing to use adequate contraceptive methods.

Other protocol-defined criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2024-09-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (safety and tolerability) | From Day 1 to Day 140
  Safety and tolerability based on the safety assessments (clinical safety laboratory tests, vital signs, weight, blood closure time and ECG parameters)
Number of participants with anti-drug antibodies | From Day 1 to Day 140
Cmax: maximum observed plasma concentration of Lu AF82422 | From Day 1 to Day 140
Tmax: time to maximum observed concentration of Lu AF82422 | From Day 1 to Day 140
AUC0-t: area under the concentration-time curve from zero to time t of Lu AF82422 | From Day 1 to Day 140
AUCinf: area under the concentration-time curve from zero to infinity of Lu AF82422 | From Day 1 to Day 140
AUC%extr: percent extrapolated AUC of total AUC0-inf of Lu AF82422 | From Day 1 to Day 140
AUMC0-inf: area under the first moment concentration-time curve from zero to infinity of Lu AF82422 | From Day 1 to Day 140
t1/2: apparent terminal elimination half-life of Lu AF82422 | From Day 1 to Day 140
MRT: mean residence time of Lu AF82422 | From Day 1 to Day 140
CL: systemic clearance of Lu AF82422 | From Day 1 to Day 140
t1/2eff: effective elimination half-life of Lu AF82422 | From Day 1 to Day 140
Vz: apparent volume of distribution of Lu AF82422 | From Day 1 to Day 140
Vss: steady-state volume of distribution of Lu AF82422 | From Day 1 to Day 140

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — H. Lundbeck A/S
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, China